CLINICAL TRIAL: NCT01248208
Title: Flu Vaccine in Egg-allergic Patients Minimizing Injections Safety Trial
Brief Title: FluMist in Egg Allergic Patients
Acronym: FluEMIST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: University of Texas (Other); University of South Alabama (Other); University of Michigan (Other); Scripps Clinic (Other)
Responsible Party: Principal Investigator, Susan Laubach, Allergy & Immunology faculty, Walter Reed Army Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 357349
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Egg Allergy; Eligible for Vaccination Against Influenza
Keywords: egg allergy; influenza vaccine
MeSH Terms: conditions — Egg Hypersensitivity; Influenza, Human | interventions — Influenza Vaccines; fluarix; FluLaval; Afluria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FluMist (LAIV) group (Experimental): FluMist influenza vaccine 0.2 mL intranasal vaccine once
  Interventions: Biological: FluMist intranasal influenza vaccine
- Flu shot (TIV) group (Active Comparator): Patients 6 months to 2 yrs or > 49 years or WITH a history of asthma symptoms / treatment within the past 12 months will receive intramuscular influenza vaccination. History/Treatment of asthma in the past 12 months is defined as follows:
  1. wheezing in the past 12 months
  2. use of inhaled corticosteroids (ICS), combined ICS / long acting beta agonist (LABA), or oral steroid in the past 12 months
  3. emergency room or acute care visit or hospitalization for asthma or wheezing in the past 12 months.
  Interventions: Biological: Intramuscular influenza injection ("flu shot")

INTERVENTIONS:
Biological: FluMist intranasal influenza vaccine — FluMist intranasal vaccine 0.2 mL will be given 0.1 mL in each nostril per manufacturer's instructions.
  Arms: FluMist (LAIV) group
Biological: Intramuscular influenza injection ("flu shot") — Subjects < 2 years or > 49 years or those with asthma symptoms or treatment within the past year will receive the intramuscular flu shot in a single injection.
  Age 6-36 months: 0.25 mL IM x 1; Age >36 months: 0.5 mL IM x 1 Boosters: All children aged 6 months-8 years who receive a seasonal influenza vaccine for the first time should be administered 2 doses. Children aged 6 months-8 years who received a seasonal vaccine for the first time during 2009-2010 but who received only 1 dose should receive 2 doses, rather than 1, during 2010-2011. In addition, for the 2010-11 influenza season, children aged 6 months-8 years who did not receive at least 1 dose of an influenza A (H1N1) 2009 monovalent vaccine should receive 2 doses of a 2010-11 seasonal influenza vaccine, regardless of previous influenza vaccination history. For all children, the second dose of a recommended 2-dose series should be administered 4 or more weeks after the initial dose.
  Other Names: Fluzone (approved for children down to 6 months); Fluvirin (age 4y and older); Agriflu (age 18y and older); Fluarix (age 3y and older); FluLaval (age 18y and older); Afluria (age 9y and older)
  Arms: Flu shot (TIV) group

SUMMARY:
With the growing public health concerns of seasonal influenza and H1N1 in the United States, the primary means by which this can be addressed is with prevention, namely, vaccination against the influenza virus. The only individuals not able to receive this vaccination in the primary care provider's office are those patients with egg allergies and, in rare circumstances, individuals with allergies to other components of the vaccine. Current guidelines allow for the administration of the influenza vaccine to patients with egg allergy using vaccines with low egg protein (ovalbumin) content or by using skin testing followed by a 5-dose desensitization protocol. Since this is impractical to perform in the primary care office and cumbersome for allergists, many egg-allergic patients simply do not receive the influenza vaccine, leaving them more vulnerable to the disease and more likely to become a source of contagion.

Several studies have suggested that influenza vaccination using a 1-2 dose protocol may be safe. This fact is due in large part to the low ovalbumin (egg protein) content in modern influenza vaccines. All studies of influenza vaccination in egg-allergic patients have been done using intramuscular trivalent inactivated influenza vaccine (TIV). However, the trivalent live-attenuated, cold-adapted influenza vaccine (LAIV), which is delivered intranasally, has a lower published ovalbumin content than the injectable vaccines, suggesting that it may also be well-tolerated by egg-allergic patients. According to several studies, LAIV may be more efficacious than TIV in children.

It is the goal of the investigators to evaluate the safety of immunizing egg-allergic individuals with the LAIV.

DETAILED DESCRIPTION:
Patients with egg allergy will be recruited into the study. Since the trivalent live-attenuated, cold-adapted influenza vaccine (LAIV) contains the lowest amount of egg protein of all available influenza vaccines on the market, those who are eligible to receive the intranasal formulation (LAIV group) (ie age 2-49y, not asthmatic) will receive FluMist; others will receive the intramuscular injection in a single dose without skin testing (TIV group). All subjects will be monitored for 30 minutes post-vaccine for any signs/symptoms of an immediate allergic reaction. Subjects will also be followed-up by phone 24-48 hours after administration to assess for any delayed allergic reaction. Data will be collected for one entire Influenza season (2010-2011).

ELIGIBILITY:
Inclusion Criteria:

* Age > 6 months
* Clinical history of allergic symptoms (hives, swelling, vomiting, respiratory problems, low blood pressure) within 2 hours after ingestion of egg OR Eczema/atopic dermatitis worsened by egg exposure
* Confirmation of clinical history by positive egg skin prick test or serum egg-specific IgE or a positive oral food challenge. [The >95% positive predictive values of egg serum IgE in subjects >2 years old with atopic dermatitis is 6 kU/L or greater. In subjects >2 years old without atopic dermatitis, the value is 7 kU/L or greater. In subjects less than 2 years old, the value is 2 kU/L or greater.]
* FluMist (LAIV) cohort: Patients age 2-49 years WITHOUT a history of asthma symptoms or treatment within the past 12 months will receive intranasal FluMist.
* Flu Shot (TIV) Intramuscular influenza vaccine cohort: Patients 6 months to 2 yrs or > 49 years or WITH a history of asthma symptoms / treatment within the past 12 months. History/Treatment of asthma in the past 12 months is defined as follows:

  1. wheezing in the past 12 months
  2. use of inhaled corticosteroids (ICS), combined ICS / long acting beta agonist (LABA), or oral steroid in the past 12 months
  3. emergency room or acute care visit or hospitalization for asthma or wheezing in the past 12 months.

Exclusion Criteria:

* Subjects who potentially have outgrown their egg allergy (no allergic reaction with ingestion of whole egg in the past 18 months and an egg serum specific IgE level ≤2 kU/L).
* Pregnancy
* Current moderate to severe illness with a fever.
* Allergy to other components of the vaccine - gentamicin, gelatin, arginine, thimerosal - or a history of a previous allergic reaction to the influenza vaccine.
* Abnormal Vital Signs.
* History of Guillain-Barre' Syndrome (GBS).
* HIV/AIDS or another disease that affects the immune system, or cancer.
* Long term health problems that are contraindicated for the LAIV or TIV.
* Receipt of a live viral vaccine within the month prior (e.g. FluMist, MMR, yellow fever, chicken pox, rotavirus, smallpox).
* Current use of any prescription medicine (e.g. antiviral) to prevent or treat influenza. (only excludes use of LAIV, may still receive TIV)
* Concurrent use of aspirin or aspirin-containing therapy in children and adolescents (2-18 years of age)(only excludes use of LAIV, may still receive TIV)
* Living with or having close contact with someone whose immune system is severely compromised (e.g. transplant recipient). (only excludes use of LAIV, may still receive TIV) Breastfeeding mothers may still receive either LAIV or TIV.
* The following medications can interfere with signs of an allergic reaction or complicate the treatment of an allergic reaction and should be discontinued as outlined below:

  1. H1 antihistamines or doxepin should be discontinued for 7 days, and diphenhydramine for 72 hrs prior.
  2. H2 antihistamines should be discontinued for 24 hrs prior.
  3. Tricyclic antidepressants should be discontinued, after consultation with the prescribing physician, for 6 weeks prior.
  4. Beta blockers should be discontinued, after consultation with the prescribing physician, for 24 hours prior.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To estimate the safety of LAIV in egg-allergic patients receiving the LAIV. | within 48 hours after vaccine administration

SECONDARY OUTCOMES:
To estimate the safety of a single, full-strength dose of TIV in egg allergic patients. | Within 48 hours of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Susan Laubach, MD, Study Director — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- See also: CDC Information on Seasonal Influenza — http://www.cdc.gov/flu/index.htm
- See also: Food Allergy and Anaphylaxis Network — http://www.foodallergy.org